CLINICAL TRIAL: NCT03376815
Title: Tumor Landscape Pathological Diagnosis by Large Tissue Sections
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2017-113R
Record Dates: First submitted 2017-11-09; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Pathology
Keywords: Tumor ,landscape ,pathological diagnosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (20):
- prostate ,traditional sample method: Samples from 100 patients with prostate carcinoma were obtained by traditional sampling method
- prostate ,landscape sample method: Samples from 100 patients with prostate carcinoma were obtained by landscape sampling method to testify the clinical value and significance of tumor landscape pathological diagnosis .
  Interventions: Diagnostic Test: landscape sample method
- liver, traditional sample method: Samples from 100 patients with liver cancer were obtained by traditional sampling method.
- liver,landscape sample method: Samples from 100 patients with liver cancer were obtained by landscape sampling method to testify the clinical value and significance of tumor landscape pathological diagnosis .
  Interventions: Diagnostic Test: landscape sample method
- esophageal ,traditional sample method: Samples from 100 patients with esophageal carcinoma were obtained by traditional sampling method.
- esophageal ,landscape sample method: Samples from 100 patients with esophageal carcinoma were obtained by landscape sampling method to testify the clinical value and significance of tumor landscape pathological diagnosis .
  Interventions: Diagnostic Test: landscape sample method
- GIST,traditional sample method: Samples from 100 patients with gastrointestinal stromal tumor were obtained by traditional sampling method.
- GIST,landscape sample method: Samples from 100 patients with gastrointestinal stromal tumor were obtained by landscape sampling method to testify the clinical value and significance of tumor landscape pathological diagnosis .
  Interventions: Diagnostic Test: landscape sample method
- colorectal ,traditional sample method: Samples from 100 patients with colorectal carcinoma were obtained by traditional sampling method.
- colorectal ,landscape sample method: Samples from 100 patients with colorectal carcinoma were obtained by landscape sampling method to testify the clinical value and significance of tumor landscape pathological diagnosis .
  Interventions: Diagnostic Test: landscape sample method
- pancreatic ,traditional sample method: Samples from 100 patients with pancreatic carcinoma were obtained by traditional sampling method.
- pancreatic,landscape sample method: Samples from 100 patients with pancreatic carcinoma were obtained by landscape sampling method to testify the clinical value and significance of tumor landscape pathological diagnosis .
  Interventions: Diagnostic Test: landscape sample method
- lung cancer,traditional sample method: Samples from 100 patients with lung cancer were obtained by traditional sampling method.
- lung cancer,landscape sample method: Samples from 100 patients with lung cancer were obtained by landscape sampling method to testify the clinical value and significance of tumor landscape pathological diagnosis .
  Interventions: Diagnostic Test: landscape sample method
- Renal ,traditional sample method: Samples from 100 patients with renal carcinoma were obtained by traditional sampling method.
- Renal carcinoma,landscape sample method: Samples from 100 patients with renal carcinoma were obtained by landscape sampling method to testify the clinical value and significance of tumor landscape pathological diagnosis .
  Interventions: Diagnostic Test: landscape sample method
- Breast cancer,traditional sample method: Samples from 100 patients with breast cancer were obtained by traditional sampling method.
- Breast cancer,landscape sample method: Samples from 100 patients with breast cancer were obtained by landscape sampling method to testify the clinical value and significance of tumor landscape pathological diagnosis .
  Interventions: Diagnostic Test: landscape sample method
- cervical ,traditional sample method: Samples from 100 patients with cervical carcinoma were obtained by traditional sampling method.
- cervical ,landscape sample method: Samples from 100 patients with cervical carcinoma were obtained by landscape sampling method to testify the clinical value and significance of tumor landscape pathological diagnosis .
  Interventions: Diagnostic Test: landscape sample method

INTERVENTIONS:
Diagnostic Test: landscape sample method — 200 cases of different tumor tissues will be compared by traditional sample method and landscape sample method to testify the clinical value and significance of tumor landscape pathological diagnosis .
  Other Names: traditional sample method
  Groups: Breast cancer,landscape sample method; GIST,landscape sample method; Renal carcinoma,landscape sample method; cervical ,landscape sample method; colorectal ,landscape sample method; esophageal ,landscape sample method; liver,landscape sample method; lung cancer,landscape sample method; pancreatic,landscape sample method; prostate ,landscape sample method

SUMMARY:
The aim of this study is to establish large tissue sections for 10 kinds of tumors. in order to observe the tumor landscape on microscope. The tumors including esophageal carcinoma,gastric carcinoma,hepatocellular carcinoma etc.200 cases of each tumor will be compared by traditional sample method and landscape sample method to testify the clinical value and significance of tumor landscape pathological diagnosis .

ELIGIBILITY:
Inclusion Criteria:

1. Older than 15-year-old
2. Did not receive preoperative preoperative chemotherapy or radiotherapy

Exclusion Criteria:

patients undergoing preoperative chemotherapy or radiotherapy

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: ZhongShan Hospital，FuDan University
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Prostate，traditional and landscape sample method | 1st January, 2018 ~30th June, 2018
  200 cases of prostate carcinoma sampled by traditional method and landscape method will be compared for precise and comprehensive pathological analysis.
liver,traditional and landscape sample method | 1st January, 2018 ~30th June, 2018
  200 cases of liver cancer sampled by traditional method and landscape method will be compared for precise and comprehensive pathological analysis.
esophageal,traditional and landscape sample method | 1st January, 2018 ~30th June, 2018
  200 cases of esophageal carcinoma sampled by traditional method and landscape method will be compared for precise and comprehensive pathological analysis.
GIST,traditional and landscape sample method | 1st July, 2018 ~31st December, 2018
  200 cases of gastrointestinal stromal tumor (GIST)sampled by traditional method and landscape method will be compared for precise and comprehensive pathological analysis.
colorectal,traditional and landscape sample method | 1st July, 2018 ~31st December, 2018
  200 cases of colorectal carcinoma sampled by traditional method and landscape method will be compared for precise and comprehensive pathological analysis.
pancreatic,traditional and landscape sample method | 1st July, 2018 ~31st December, 2018
  200 cases of pancreatic carcinoma sampled by traditional method and landscape method will be compared for precise and comprehensive pathological analysis.
lung, traditional and landscape sample method | 1st July, 2018 ~31st December, 2018
  200 cases of lung cancer sampled by traditional method and landscape method will be compared for precise and comprehensive pathological analysis.
renal,traditional and landscape sample method | 1st July, 2018 ~31st December, 2018
  200 cases of renal carcinoma sampled by traditional method and landscape method will be compared for precise and comprehensive pathological analysis.
breast,traditional and landscape sample method | 1st July, 2018 ~31st December, 2018
  200 cases of breast cancer sampled by traditional method and landscape method will be compared for precise and comprehensive pathological analysis.
cervical,traditional and landscape sample method | 1st July, 2018 ~31st December, 2018
  200 cases of cervical carcinoma sampled by traditional method and landscape method will be compared for precise and comprehensive pathological analysis.